CLINICAL TRIAL: NCT06700226
Title: AblaView® Unipolar PFA OCR-guided Feasibility Study - First in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medlumics (Industry)
Collaborators: Clinical Accelerator (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 48437
Record Dates: First submitted 2024-11-14; First posted 2024-11-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal AF
Keywords: Atrial Fibrillation; PFA; Optically guided
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single-center, open, single-arm, exploratory clinical investigation. This clinical investigation will include up to 10 subjects in 1 site. All subjects treated will be followed up for 3 months or up to re-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated under PFA (Experimental): Single-Arm study, all patients included will undergo PFA using AblaView® Unipolar PFA System
  Interventions: Device: AblaView® Unipolar PFA System

INTERVENTIONS:
Device: AblaView® Unipolar PFA System — Patients with symptomatic paroxysmal atrial fibrillation will be treated with the AblaView® Unipolar PFA System system to achieve electrical isolation of the pulmonary veins. The AblaView® Unipolar PFA Catheter is a regular PFA irrigated catheter. The tip of the catheter has 7 holes distributed around that deliver at the same time irrigation and near infrared light for the OCR system, which will be processed and interpreted by the Console.

SUMMARY:
Exploratory Clinical Investigation to evaluate the feasibility and safety of the AblaView® Unipolar Percutaneous Ablation Irrigated Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation using Polarization Sensitive Optical Coherence Reflectometry (PS-OCR) to guide delivery of Pulsed Field Ablation (PFA) lesions - First in Man

DETAILED DESCRIPTION:
Exploratory Clinical Investigation to evaluate the feasibility and safety of the AblaView® Unipolar Percutaneous Ablation Irrigated Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation using Polarization Sensitive Optical Coherence Reflectometry (PS-OCR) to guide delivery of Pulsed Field Ablation (PFA) lesions - First in Man

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the following criteria:

1. Symptomatic Paroxysmal Atrial Fibrillation (PAF) with at least one documented episode in the 6 previous months (according to the ESC 2020 guidelines and AHA/ACC 2023 Guidelines). Documentation may include ECG, trans-telephonic monitor (TTM), Holter monitor (HM), or telemetry strips.
2. Eligible for de novo catheter intra-atrial ablation (e.g., pulmonary vein isolation).
3. Eligible for Transesophageal echocardiography (TEE) or Intracardiac Echocardiography (ICE) (AHA/ACC/HRS 2014 Guidelines for AF Management pertaining to anticoagulation at the time of cardioversion and the update in 2023) performed within 24 hours of the ablation procedure in all patients with AF of 48 hours duration or of unknown duration if adequate systemic anticoagulation has not been maintained for at least 1 month prior to AF ablation.
4. Antero-posterior left atrial diameter ≤ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT) within 3 months prior to the procedure.
5. Age ≥ 18 years and ≤ 85 years on the day of enrollment.
6. Voluntarily accepts participation after being duly informed of the ablation procedure and its risks, as well as the remapping procedure planned three months later, by signing the informed consent form.

Exclusion Criteria:

1. Persistent or long-standing persistent AF.
2. Arrhythmia due to reversible causes, including thyroid disorders, acute alcohol intoxication, electrolyte disorders, and other major surgical procedures in the preceding three months.
3. Myocardial infarction (MI), acute coronary syndrome percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within the preceding 3 months.
4. Antero-posterior Left atrial diameter > 5.5 cm
5. Previous left atrial ablation procedures, either surgical or catheter ablation.
6. Prior left atrial intervention, surgical procedure, or incision with resulting scar, including AF ablation or LAA closure.
7. Previous tricuspid or mitral valve replacement or repair.
8. Presence of an implantable cardiac defibrillator (ICD).
9. Heart disease for which corrective surgery is anticipated within 6 months.
10. Active systemic infection.
11. Bleeding diathesis or suspected procoagulant state.
12. Contraindication to long-term antithromboembolic therapy.
13. Presence of a condition that precludes appropriate vascular access.
14. Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73 m2 or has ever received dialysis renal failure requiring dialysis.
15. Body mass index > 40.
16. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with premedication.
17. Contraindication to general anesthesia (GA)
18. Contraindications to computed tomography.
19. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms.
20. Positive pregnancy test results for female subjects with childbearing potential.
21. Has known pulmonary vein stenosis, or other anatomic or concomitant conditions that, in the investigator's opinion, could limit the subject's ability to participate in the study, comply with follow-up requirements, or impact the scientific soundness of the study results.
22. In the opinion of the Principal Investigator (PI), it is unlikely to survive the clinical investigation plan with a follow-up period of twelve months.
23. Clinically significant psychological conditions that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
24. Currently participating in another clinical investigation or participating in a clinical investigation that may interfere with this clinical investigation within 30 days prior to screening.
25. Severely compromised LVEF (LVEF <40%)
26. The presence of intracardiac thrombus (e.g., LA), myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
27. Severe mitral regurgitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Realtime predictability of PFA ablation lesion chronicity | Up to 3 months
  Feasibility:
  3-month Validation: Predictability Assessment by PS-OCR and PFA Lesions continuity and chronicity at 3-month remapping. Evaluation of the predictability of chronicity of ablation lesions in terms of Accuracy, Specificity and Sensitivity
Safety Acute | Up to 3 months
  Serious procedure- and device-related adverse events. Serious adverse events, and their relatedness to the AblaView Unipolar PFA System or procedure will be adjudicated by the Clinical Events Committee. The sites are required to report all adverse events.

SECONDARY OUTCOMES:
Procedure Parameters | The day of the procedure
  * Skin-to-skin procedural time, minutes
  * Device left atrial dwell time, minutes
  * Time between first and last application, minutes
  * Fluoroscopy time during procedure, minutes
  * Total amount of PFA energy delivered in, joules.
  * Number of applications per targeted vein and/or isolation and for complete procedure, number
Per procedure (Ablation/remapping) optical parameters | The day of procedure
  * Detection of optical signals to evaluate contact and birefringence in the left atria, yes or no
  * Detection and quantification of changes in birefringence during ablation, in %
  * Detection of gaps in the continuous ablation/isolation lines during ablation procedure, yes or no
Procedure Validation | The day of the procedure
  Acute Validation (20 to 30) min at least after the completion of each line/isolation by Electrical and optical isolation of targeted pulmonary veins (PVs), yes or no
Recurrence | Up to 3 months
  Recurrence or new occurrence of arrhythmias controlled by Holter 48-hrs and by TTM weekly and triggered by symptoms.
Improvement in the Quality of Life | At 3 months
  * Atrial Fibrillation Effect on Quality-of-Life (AFEQT) score difference between baseline and at 3 month
  * European Quality of Life-5 Dimensions (EQ-5D-5L) score difference between baseline and at 3 month in total and for mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Safety at 1 month | At 1 month
  MACE (30d)
Safety at 3 months | Between 1 month and 3 months
  Occurence of Atrial/Ventricular Arrhythmias, Stroke, HF

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, PhD, Study Chair — Division of Cardiology, McGill University Health Centre, McGill University, Montreal, Quebec, Canada; Raphael Martins, MD, PhD, Study Chair — University of Rennes, CHU Rennes, Rennes, France; Askar Sabirov, MD, Principal Investigator — Cardiology Department, AKFA Medline University Hospital, Tashkent, Uzbekistan; Giorgi Papiashvili, MD, PhD, Study Chair — Israeli-Georgian Medical Research Clinic Healthycore and European University, Tbilisi; Georgia.
Locations (1):
- Ezgu Niyat, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
Small feasibility studies of device products